CLINICAL TRIAL: NCT01595061
Title: A Phase II Trial Evaluating Cisplatin (NSC #119875) and Gemcitabine (NSC #613327) Concurrent With Intensity-Modulated Radiation Therapy (IMRT) in the Treatment of Locally Advanced Squamous Cell Carcinoma of the Vulva (NCT #01595061)
Brief Title: Radiation Therapy, Gemcitabine Hydrochloride, and Cisplatin in Treating Patients With Locally Advanced Squamous Cell Cancer of the Vulva
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0279; NCI-2012-01964 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000732793; GOG-0279 (Other: NRG Oncology); GOG-0279 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Stage III Vulvar Cancer AJCC v7; Stage IIIA Vulvar Cancer AJCC v7; Stage IIIB Vulvar Cancer AJCC v7; Stage IIIC Vulvar Cancer AJCC v7; Stage IVA Vulvar Cancer AJCC v7; Vulvar Squamous Cell Carcinoma
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (IMRT, gemcitabine, cisplatin, surgery) (Experimental): Patients undergo IMRT 5 days a week for 6 weeks. Patients also receive gemcitabine hydrochloride IV over 30 minutes and cisplatin IV over 60 minutes weekly for 6 weeks in the absence of disease progression or unacceptable toxicity. Within 6-8 weeks after completion of chemoradiation patients undergo local core biopsy to confirm response or surgical excision of gross residual disease in the vulva and/or inguinal-femoral lymph nodes.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Therapeutic Conventional Surgery — Undergo local core biopsy or surgical excision

SUMMARY:
This phase II trial studies how well radiation therapy works when given with gemcitabine hydrochloride and cisplatin work in treating patients with squamous cell cancer of the vulva that has spread from where it started to nearby tissue or lymph nodes. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving radiation therapy together with gemcitabine hydrochloride and cisplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of cisplatin, gemcitabine (gemcitabine hydrochloride), and intensity-modulated radiation therapy (IMRT) in achieving a complete pathologic response when used for the primary treatment of locally-advanced squamous cell carcinoma of the vulva.

SECONDARY OBJECTIVES:

I. To determine the efficacy of cisplatin, gemcitabine, and IMRT in achieving a complete clinical response when used for the primary treatment of locally-advanced squamous cell carcinoma of the vulva.

II. To determine the vulvar progression-free survival and groin progression-free survival in women treated with cisplatin, gemcitabine and IMRT for locally advanced vulvar carcinoma.

III. To determine the toxicity and surgical morbidity of the combined modality approach of cisplatin, gemcitabine and IMRT followed by reduced-scope surgery for the treatment of locally-advanced vulvar carcinoma.

OUTLINE:

Patients undergo IMRT 5 days a week for 6 weeks. Patients also receive gemcitabine hydrochloride intravenously (IV) over 30 minutes and cisplatin IV over 60 minutes weekly for 6 weeks in the absence of disease progression or unacceptable toxicity. Within 6-8 weeks after completion of chemoradiation patients undergo local core biopsy to confirm response or surgical excision of gross residual disease in the vulva and/or inguinal-femoral lymph nodes.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced, previously untreated squamous cell carcinoma of the vulva
* Patients with T2 or T3 primary tumors (N0-3, M0) not amenable to surgical resection by standard radical vulvectomy
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets >= 100,000/mcl
* Creatinine =< 1.5 times institutional upper limit of normal (ULN) OR calculated creatinine clearance >= 60 mL/min
* Bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 x ULN
* Alkaline phosphatase =< 3 x ULN
* Patients judged capable of tolerating a radical course of chemoradiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III protocol or Rare Tumor protocol for the same patient population
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients with a GOG performance status of 0, 1, or 2

Exclusion Criteria:

* Patients with recurrent carcinoma of the vulva regardless of previous treatment
* Patients who have received prior pelvic radiation or cytotoxic chemotherapy
* Patients with vulvar melanomas or sarcomas
* Patients with circumstances that will not permit completion of the study or the required follow-up
* Patients with evidence of active septicemia, severe infection, gastrointestinal bleeding or severe gastrointestinal symptoms requiring medical or surgical therapy
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2022-09-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Neil S Horowitz, Principal Investigator — NRG Oncology
Locations (193):
- United States (193):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Women's Cancer Care Associates LLC, Albany, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Derived] Horowitz NS, Deng W, Peterson I, Mannel RS, Thompson S, Lokich E, Myers T, Hanjani P, O'Malley DM, Chung KY, Miller DS, Ueland FR, Dizon DS, Miller A, Mayadev JS, Leath CA 3rd, Monk BJ. Phase II Trial of Cisplatin, Gemcitabine, and Intensity-Modulated Radiation Therapy for Locally Advanced Vulvar Squamous Cell Carcinoma: NRG Oncology/GOG Study 279. J Clin Oncol. 2024 Jun 1;42(16):1914-1921. doi: 10.1200/JCO.23.02235. Epub 2024 Apr 4. PMID 38574312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: GOG-0279 was activated on 07/02/2012 and closed to accrual on February 20, 2020.
Groups:
- GEM+CIS+IMRT: Gemcitabine 50 mg/m2 and Cisplatin 40mg/m2 administered weekly throughout IMRT radiation therapy. Gemcitabine will be infused prior to cisplatin and given over approximately 30 minutes while the cisplatin will be delivered over approximately 60 minutes.
Period: Overall Study
Arm/Group | GEM+CIS+IMRT
Started | 57
Completed | 53
Not Completed | 4
Not completed — Never Treated | 3
Not completed — Inadequate Pathology | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated
Arm/Group | GEM+CIS+IMRT
Number analyzed (Participants) | 53
Age, Customized [Count of Participants; unit: Participants]
  20 - 29 years | 1
  30 - 39 years | 0
  40 - 49 years | 6
  50 - 59 years | 23
  60 - 69 years | 10
  70 - 79 years | 8
  >= 80 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 50
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response
Description: Percentage of participants with complete pathologic response. Complete pathologic response is defined as negative local core biopsy or FNA specimens following primary chemo-radiation therapy.
Time Frame: 6 -8 weeks after completion of chemo-radiation
Population: Eligible and treated
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GEM+CIS+IMRT
Number analyzed (Participants) | 53
percentage of participants | 73.6 [64 to 100]

2. Secondary Outcome: Complete Clinical Response
Description: Percentage of participants with complete clinical response. Complete clinical response is defined as no clinical/radiographic evidence of primary disease (vulva or groin) following primary chemo-radiation therapy.
Time Frame: 6-8 weeks after completion of chemo-radiation
Population: Eligible and Treated
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GEM+CIS+IMRT
Number analyzed (Participants) | 53
percentage of participants | 71.7 [60 to 82]

3. Secondary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: During treatment period and up to 30 days after stopping the study treatment. The median for duration of study treatment was 2.1 months with a range from 1.2 months to 4.6 months.
Population: Eligible and Treated
Measure: Count of Participants; unit: Participants
Arm/Group | GEM+CIS+IMRT
Number analyzed (Participants) | 53
Participants
  Leukopenia | 27
  Thrombocytopenia | 20
  Neutropenia | 20
  Anemia | 20
  Other Investigations | 7
  Other blood and lymphatic disorders | 8
  Cardiac disorders | 2
  Gastrointestinal disorders | 10
  General disorders and administration site conditions | 5
  Infections and infestations | 5
  Injury, poisoning and procedural complications | 20
  Metabolism and nutrition disorders | 19
  Musculoskeletal and connective tissue disorders | 2
  Peripheral sensory neuropathy | 1
  Other nervous system disorders | 2
  Renal and urinary disorders | 1
  Reproductive system and breast disorders | 7
  Respiratory, thoracic and mediastinal disorders | 1
  Skin and subcutaneous tissue disorders | 4
  Surgical and medical procedures | 1
  Vascular disorders | 5

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Estimate for probability of progression free survival by Kaplan-Meier method, where progression-free survival is defined as the period of time from study entry to time of disease progression, death or date of last contact, whichever occurs first. PFS is censored in patients who are alive and have not progressed. Progression is assessed by RECIST 1.1
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first. The median for observed PFS was 26.2 month with a range from 1.5 months to 82.4 months
Population: Eligible and treated
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GEM+CIS+IMRT
Number analyzed (Participants) | 53
percentage of participants | 75 [63 to 83]

ADVERSE EVENTS:
Time Frame: During treatment period and up to 30 days after stopping the study treatment. The median for duration of study treatment was 2.1 months with a range from 1.2 months to 4.6 months.
Arm/Group | GEM+CIS+IMRT
All-Cause Mortality (participants affected / at risk) | 1/53
Serious Adverse Events (participants affected / at risk) | 24/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEM+CIS+IMRT (N=53)
Anemia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Ventricular Tachycardia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Sudden Death Nos (General disorders) | 1
Skin Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Vascular Access Complication (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Platelet Count Decreased (Investigations) | 2
Lymphocyte Count Decreased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Seizure (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEM+CIS+IMRT (N=53)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 42
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Atrial Fibrillation (Cardiac disorders) | 2
Mobitz Type I (Cardiac disorders) | 1
Supraventricular Tachycardia (Cardiac disorders) | 1
Sinus Bradycardia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 3
Sinus Tachycardia (Cardiac disorders) | 5
Chest Pain - Cardiac (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 4
Blurred Vision (Eye disorders) | 2
Floaters (Eye disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 20
Diarrhea (Gastrointestinal disorders) | 39
Vomiting (Gastrointestinal disorders) | 21
Bloating (Gastrointestinal disorders) | 2
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 5
Proctitis (Gastrointestinal disorders) | 3
Mucositis Oral (Gastrointestinal disorders) | 2
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 3
Anal Pain (Gastrointestinal disorders) | 3
Gingival Pain (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 38
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Rectal Pain (Gastrointestinal disorders) | 2
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 1
General Disorders And Administration Site Conditio (General disorders) | 5
Pain (General disorders) | 9
Malaise (General disorders) | 2
Localized Edema (General disorders) | 3
Non-Cardiac Chest Pain (General disorders) | 2
Edema Limbs (General disorders) | 12
Fatigue (General disorders) | 42
Fever (General disorders) | 6
Chills (General disorders) | 2
Allergic Reaction (Immune system disorders) | 1
Infections And Infestations - Other (Infections and infestations) | 5
Vulval Infection (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Hepatitis Viral (Infections and infestations) | 1
Vaginal Infection (Infections and infestations) | 4
Urinary Tract Infection (Infections and infestations) | 13
Vascular Access Complication (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Dermatitis Radiation (Injury, poisoning and procedural complications) | 35
Burn (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Investigations - Other (Investigations) | 2
Weight Loss (Investigations) | 5
Platelet Count Decreased (Investigations) | 38
Lymphocyte Count Decreased (Investigations) | 7
Creatinine Increased (Investigations) | 8
Neutrophil Count Decreased (Investigations) | 31
Blood Bilirubin Increased (Investigations) | 1
White Blood Cell Decreased (Investigations) | 41
Aspartate Aminotransferase Increased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 6
Alanine Aminotransferase Increased (Investigations) | 4
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 25
Hypokalemia (Metabolism and nutrition disorders) | 19
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 18
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypercalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 17
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Seizure (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 7
Paresthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Cognitive Disturbance (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 6
Delirium (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Urine Discoloration (Renal and urinary disorders) | 1
Urinary Urgency (Renal and urinary disorders) | 5
Urinary Tract Obstruction (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 3
Urinary Incontinence (Renal and urinary disorders) | 7
Urinary Tract Pain (Renal and urinary disorders) | 12
Urinary Frequency (Renal and urinary disorders) | 15
Proteinuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 4
Cystitis Noninfective (Renal and urinary disorders) | 2
Chronic Kidney Disease (Renal and urinary disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 3
Vaginal Pain (Reproductive system and breast disorders) | 11
Vaginal Hemorrhage (Reproductive system and breast disorders) | 7
Perineal Pain (Reproductive system and breast disorders) | 8
Pelvic Pain (Reproductive system and breast disorders) | 5
Vaginal Discharge (Reproductive system and breast disorders) | 9
Vaginal Inflammation (Reproductive system and breast disorders) | 1
Genital Edema (Reproductive system and breast disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 6
Skin Ulceration (Skin and subcutaneous tissue disorders) | 3
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6
Pain Of Skin (Skin and subcutaneous tissue disorders) | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1
Thromboembolic Event (Vascular disorders) | 6
Superficial Thrombophlebitis (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 8
Hot Flashes (Vascular disorders) | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT01595061/Prot_SAP_000.pdf